CLINICAL TRIAL: NCT02692781
Title: A Phase I, Randomized, Single-Blinded, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of MOD-6031 in Healthy Volunteers
Brief Title: A Single-dose, Dose-escalation Study of a Long-acting MOD-6031 in Healthy Overweight or Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-6-001
Record Dates: First submitted 2016-02-04; First posted 2016-02-26 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- Dose Cohort 1 (Experimental): 20mg MOD-6031 / Placebo
  Interventions: Drug: MOD-6031; Other: Placebo control
- Dose Cohort 2 (Experimental): 50mg MOD-6031 / Placebo
  Interventions: Drug: MOD-6031; Other: Placebo control
- Dose Cohort 3 (Experimental): 100mg MOD-6031 / Placebo
  Interventions: Drug: MOD-6031; Other: Placebo control
- Dose Cohort 4 (Experimental): 150mg MOD-6031 / Placebo
  Interventions: Drug: MOD-6031; Other: Placebo control
- Dose Cohort 5 (Experimental): 200mg MOD-6031 / Placebo
  Interventions: Drug: MOD-6031; Other: Placebo control

INTERVENTIONS:
Drug: MOD-6031
Other: Placebo control

SUMMARY:
MOD-6031 is a long-acting reversibly PEGylated oxyntomodulin (OXM) therapeutic. The active moiety is a gastrointestinal neuropeptide with a sequence identical to endogenous human OXM and is an agonist for both glucagon-like peptide-1 (GLP1) and glucagon (GCG) receptors. The peptide is a natural appetite suppressant, secreted by L-cells in the digestive system following food intake leading to a decrease in gastric emptying, satiety after crossing the blood-brain barrier, and regulation of insulin and glucose levels. Thus, MOD-6031 is being developed as a treatment for high risk subjects (obese) to increase weight loss, reduce food intake and increase glycemic control.

DETAILED DESCRIPTION:
This will be a a randomized, single-blind, placebo-controlled, single-dose, dose-escalation study. Five escalating dose groups are planned, with 8 subjects per dose group, randomized in 3:1 ratio to receive a single dose of MOD-6031 or matching Placebo (6 MOD-6031 to 2 placebo subjects). The initial MOD-6031 dose will be 20 mg, followed by single doses of 50 mg, 100 mg, 150 mg and 200 mg. Each subject will receive a single study drug injection in the morning (dosing day designated as Day 0) and will be monitored for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, between 18 to 55 years of age.
* BMI 27-35 Kg/m2 (inclusive).
* Generally good health.
* Triglyceride ≤ 400mg/ml
* ECG with no clinically significant abnormalities.
* Negative HIV, hepatitis B or hepatitis C serology tests at screening
* No significant abnormalities in clinical laboratory parameters
* No history of alcohol or drug abuse.

Exclusion Criteria:

* History of clinically significant medical condition.
* Any cardiac conduction defect.
* Any acute or unstable disease.
* History of malignancy diagnosed within the past 5 years.
* Known or suspected diabetes and/or HbA1C >6.4% on screening.
* Known allergy to any drug.
* Treatment with weight loss drugs (within 3 months prior to dosing).
* Liposuction or other surgery for weight loss within the last year.
* Evidence of eating disorders (bulimia, binge eating).
* History of regular alcohol consumption exceeding.
* Use of tobacco or nicotine-containing products.
* Subjects that have difficulty fasting or consuming the standard meals that will be provided.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Composite safety and tolerability parameters as measured by adverse events, electrocardiograms (ECG), laboratory results, vital signs and injection site reactions | 30 days

SECONDARY OUTCOMES:
Cmax of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
Tmax of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
AUC(0-t) of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
AUC(inf) of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
Elimination rate constant of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
T(½) of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
CL/F of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days
Vz/F of MOD-6031 and its hydrolyzed derivatives (PEG-FMS and OXM peptide) | 0 to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel